CLINICAL TRIAL: NCT04402944
Title: Pulmozyme to Improve COVID-19 ARDS Outcomes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); South Shore Hospital (Other)
Responsible Party: Principal Investigator, Benjamiin Raby, Chief of Respiratory Diseases, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P00035140
Record Dates: First submitted 2020-05-12; First posted 2020-05-27 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: COVID
Keywords: Pulmozyme; Pneumonia; ARDS
MeSH Terms: conditions — Pneumonia | interventions — dornase alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Drug (Experimental): Study drug
  Interventions: Drug: Pulmozyme
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pulmozyme — Pulmozyme 2.5 mg BID
  Other Names: Dornase alfa
  Arms: Study Drug
Drug: Placebo — Saline 2.5 mL BID
  Arms: Placebo

SUMMARY:
This is a randomized double-blind placebo-controlled Phase II trial of recombinant human deoxyribonuclease I (rhDNase I) - Pulmozyme - in mechanically ventilated patients with COVID-19 pneumonia.

Patients admitted to the ICU with severe COVID-19 pneumonia who require mechanical ventilation will be invited to participate in this study. Potential subjects will be identified from medical record review or from direct contact with physicians. Investigators will check medical history and confirm eligibility. Informed consent will be obtained from either the patient or designated healthcare proxy.

60 subjects will be enrolled. After obtaining informed consent, patients will be randomized 2:1 to Pulmozyme 2.5 mg BID for up to 28 days or until they are no longer receiving mechanical ventilation, whichever is sooner plus standard of care vs. placebo normal saline 2.5 ml plus standard of care.

ELIGIBILITY:
Inclusion Criteria:

* ICU admission for pneumonia complicated by respiratory failure.
* RT-PCR (or equivalent) confirmed COVID-19 infection.
* Intubated and on mechanical ventilation within 120 hours of initiation of mechanical ventilation.
* Age ≥ 3 years of age.

Exclusion Criteria:

* Allergy or known intolerance to Pulmozyme or Chinese Hamster Ovary cell products
* History of moderate to severe asthma, cystic fibrosis, or severe COPD (baseline FEV1 ≤ 40% predicted)
* Active malignancy other than basal cell melanoma or in situ breast cancer
* Unstable angina
* Chronic liver disease as judged by the investigator that would pose significant risk to participation
* Chronic renal disease as judged by the investigator that would pose significant risk to participation
* Inability to obtain informed consent from patient or legally authorized representative (LAR)
* Pregnant or breastfeeding Use of extracorporeal membrane oxygenation (ECMO)
* Prisoner status
* Concurrent treatment with other inhaled investigational agent for COVID-19**
* Patient, surrogate, or physician not committed to full support (exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)
* Moribund patient not expected to survive 24 hours
* Active hemoptysis

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-05 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free days at 28 days | 28 days
  Primary outcome

SECONDARY OUTCOMES:
change in airway resistance | 28 days
  change in airway resistance
change in lung compliance | 28 days
  Change in lung compliance
oxygenation (PaO2/FiO2 ratio) | 28 days
  oxygenation
length of stay (ICU and hospital) | 28 days
  length of stay
rate of barotrauma | 28 days
  rate of batotrauma
mortality. | 28 days
  mortality

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts